CLINICAL TRIAL: NCT02801045
Title: Art Therapy in Palliative Care: Study of Identification and Understanding of the Mechanisms of Change in the Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-ART-2016-14
Record Dates: First submitted 2016-05-30; First posted 2016-06-15 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Psychological Stress; Suffering; Advanced Cancers
MeSH Terms: conditions — Stress, Psychological | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- art therapy (Experimental): Individual 30-60 minutes art therapy sessions, twice a week, offering visual arts materials.
  Interventions: Behavioral: art therapy

INTERVENTIONS:
Behavioral: art therapy — Patient's creativity is stimulated by visual arts materials and various art therapy techniques including punctual use of music, poetry and body expression. The intervention, based on the investigators previous experience, is founded on:
  * humanistic phenomenological focus
  * transpersonal therapeutic bound
  * transdisciplinarity in the artistic approach
  * integrative-relational specialized counseling of the grief, loss and trauma aspects.

SUMMARY:
This study evaluates from the patient's perspective which elements of the own artistic creative process are the source of a beneficial change for him/her and how those elements influence in their end of life experience.

DETAILED DESCRIPTION:
In previous quantitative studies about the effect of an art therapy intervention in adult cancer inpatients of the Palliative Care Unit, the investigators evidenced significant improvements in the symptom control of malaise, anxiety, depression and pain.

This study is designed to deepen the understanding of specific action mechanisms which lead to those therapeutic benefits and quality of life implications for patients with life-threatening illness in which a situation of suffering is frequently detected.

The investigators will determine from the subjective patient's experience which specific elements of the artistic creative process (including production of art and art products) may lead to changes in the symptom perception, in meaning and healing process and in the personal perspective about the end of life situation.

ELIGIBILITY:
Inclusion Criteria:

* advanced-cancer adult inpatients of the Palliative Care Unit
* informed consent

Exclusion Criteria:

* altered cognitive function (Mini-Mental Test < 24)
* physical decline (palliative care team's criteria) that impedes the art therapy process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Reflect Interview (RI) using audio recording. | After the making of a minimum of 5 art pieces, an average of 2 weeks
  An art based interview is administered and involves the patients selecting 2 significant artworks from their art therapy productions. The patient is asked by the art therapist for a narrative of how one artwork relates to the other in the context of his/her lived experience. The art therapy dialogue from the RI is transcribed and subjected to thematic analysis.

SECONDARY OUTCOMES:
Art therapy process from the art therapist perspective. | Every day of art therapy session, with an average of 2 sessions a week, over a period of 2 years.
  Detailed notes and photographical register.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pascual, MD, Principal Investigator — Palliative Care Unit, Sant Pau Hospital, Barcelona, Spain.
Locations (1):
- Hospital Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No